CLINICAL TRIAL: NCT07184606
Title: Clinical Study of the Safety and Pharmacokinetics of the Drug Fluorothiazinone (N.F. Gamaleya NRCEM), a Concentrate for Solution Preparation for Infusion With Participation of Adult Healthy Volunteers.
Brief Title: Clinical Study of the Safety and Pharmacokinetics of the Drug Fluorothiazinone, a Concentrate for Solution Preparation for Infusion.
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Gamaleya Research Institute of Epidemiology and Microbiology, Health Ministry of the Russian Federation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 08-FT-2025
Record Dates: First submitted 2025-09-18; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Safety and Pharmacokinetics
MeSH Terms: interventions — Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- ¼ of the full (target) dose (solution, 5 ml) (Experimental): 1. st cohort of volunteers: 3 healthy volunteers will receive ¼ of the full (target) dose of the study drug, and 1 healthy volunteer will receive placebo.
  2. nd cohort of volunteers: in case of AE in 1st cohort, 3 healthy volunteers will receive ¼ of the full (target) dose of the study drug.
  Interventions: Drug: ¼ of the full (target) dose (solution, 5 ml); Other: Placebo
- ½ of the full (target) dose (solution, 10 ml) (Experimental): 1. st cohort of volunteers: 3 healthy volunteers will receive ½ of the full (target) dose of the study drug, and 1 healthy volunteer will receive placebo.
  2. nd cohort of volunteers: in case of AE in 1st cohort, 3 healthy volunteers will receive ½ of the full (target) dose of the study drug.
  Interventions: Drug: ½ of the full (target) dose (solution, 10 ml); Other: Placebo
- full dose (solution, 20 ml) (Experimental): 1. st cohort of volunteers: 3 healthy volunteers will receive full (target) dose of the study drug, and 1 healthy volunteer will receive placebo.
  2. nd cohort of volunteers: in case of AE in 1st cohort, 3 healthy volunteers will receive full (target) dose of the study drug.
  Interventions: Drug: full dose (solution, 20 ml); Other: Placebo
- 1 ½ of the full (target) dose (solution, 30 ml) (Experimental): 1. st cohort of volunteers: 3 healthy volunteers will receive 1 ½ of the full (target) dose of the study drug, and 1 healthy volunteer will receive placebo.
  2. nd cohort of volunteers: in case of AE in 1st cohort, 3 healthy volunteers will receive 1 ½ of the full (target) dose of the study drug.
  Interventions: Drug: 1 ½ of the full (target) dose (solution, 30 ml); Other: Placebo
- 2 full doses (solution, 40 ml) (Experimental): 1. st cohort of volunteers: 3 healthy volunteers will receive 2 full (target) doses of the study drug, and 1 healthy volunteer will receive placebo.
  2. nd cohort of volunteers: in case of AE in 1st cohort, 3 healthy volunteers will receive 2 full (target) doses of the study drug.
  Interventions: Drug: 2 full doses (solution, 40 ml); Other: Placebo
- course administration of the selected dose (Experimental): 10 healthy volunteers will receive course administration of the selected dose, and 1 healthy volunteer will receive placebo
  Interventions: Drug: course administration of the selected dose; Other: Placebo

INTERVENTIONS:
Drug: ¼ of the full (target) dose (solution, 5 ml) — 1. st cohort of volunteers: 3 healthy volunteers will receive ¼ of the full (target) dose of the study drug, and 1 healthy volunteer will receive placebo (parenteral administration).
  2. nd cohort of volunteers: in case of AE in 1st cohort, 3 healthy volunteers will receive ¼ of the full (target) dose of the study drug (parenteral administration).
  Arms: ¼ of the full (target) dose (solution, 5 ml)
Drug: ½ of the full (target) dose (solution, 10 ml) — 1. st cohort of volunteers: 3 healthy volunteers will receive ½ of the full (target) dose of the study drug, and 1 healthy volunteer will receive placebo (parenteral administration).
  2. nd cohort of volunteers: in case of AE in 1st cohort, 3 healthy volunteers will receive ½ of the full (target) dose of the study drug (parenteral administration).
  Arms: ½ of the full (target) dose (solution, 10 ml)
Drug: full dose (solution, 20 ml) — 1. st cohort of volunteers: 3 healthy volunteers will receive full (target) dose of the study drug, and 1 healthy volunteer will receive placebo (parenteral administration).
  2. nd cohort of volunteers: in case of AE in 1st cohort, 3 healthy volunteers will receive full (target) dose of the study drug (parenteral administration).
  Arms: full dose (solution, 20 ml)
Drug: 1 ½ of the full (target) dose (solution, 30 ml) — 1. st cohort of volunteers: 3 healthy volunteers will receive 1 ½ of the full (target) dose of the study drug, and 1 healthy volunteer will receive placebo (parenteral administration).
  2. nd cohort of volunteers: in case of AE in 1st cohort, 3 healthy volunteers will receive 1 ½ of the full (target) dose of the study drug (parenteral administration).
  Arms: 1 ½ of the full (target) dose (solution, 30 ml)
Drug: 2 full doses (solution, 40 ml) — 1. st cohort of volunteers: 3 healthy volunteers will receive 2 full (target) doses of the study drug, and 1 healthy volunteer will receive placebo (parenteral administration).
  2. nd cohort of volunteers: in case of AE in 1st cohort, 3 healthy volunteers will receive 2 full (target) dose of the study drug (parenteral administration).
  Arms: 2 full doses (solution, 40 ml)
Drug: course administration of the selected dose — 10 healthy volunteers will receive course administration of the selected dose, and 1 healthy volunteer will receive placebo.
  Arms: course administration of the selected dose
Other: Placebo — 1 healthy volunteer from the 1st cohort of each group will receive placebo (parenteral administration)

SUMMARY:
A two-stage placebo-controlled open-label safety and pharmacokinetics study of the drug Fluorothiazinone, a concentrate for the preparation of an infusion solution, with participation of adult healthy volunteers.

Stage 1 - single administration; dose escalation will be carried out in sequential groups after evaluation of side effects data on day 7.

Stage 2 - course administration of the selected dose.

Total number of healthy replacement volunteers: 5.

ELIGIBILITY:
INCLUSION CRITERIA

Each potential volunteer for inclusion in the Study should meet all of the following criteria:

1. Written Informed Consent to participate in the Study.
2. The ability to understand the requirements for the study participants, and the willingness to follow the procedures provided in the Study Protocol.
3. Men and women, age limits: min.: 18, max.: 45.
4. Healthy according to the results of a medical examination: no history of pathology in the gastrointestinal tract, liver, kidneys, cardiovascular system, central nervous system, musculoskeletal system, genitourinary, immune and endocrine systems, or blood, which may affect the safety of the volunteer and the assessment of the Study results (no diseases or clinically significant abnormalities were revealed by clinical, instrumental, and laboratory tests).
5. Negative test results for HIV, hepatitis B and C, syphilis.
6. A negative urine test result for presence of narcotic and psychostimulants.
7. A negative alcohol content test.
8. Indicators of general and biochemical blood analysis at screening in reference interval: 1.1 X Lower limit - 0.9 X Upper limit.
9. No contraindications to infusion therapy.
10. A negative pregnancy test result.
11. Consent to the use effective methods of contraception during the entire period of participation in the Study.

NON-INCLUSION CRITERIA

The potential volunteer will not be included in the Study in the following cases:

1. Inability to read in Russian; inability or unwillingness to understand the essence of the Study. Any other condition that restricts the validity of obtaining informed consent or may affect the volunteer's ability to participate in the Study.
2. Acute infectious diseases within 2 weeks and non-infectious diseases, exacerbations of chronic diseases within 4 weeks before the screening.
3. Hypersensitivity to fish proteins, eggs, soy, peanut butter or the components of the drug SMOFlipid.
4. The volunteer's participation in any other study within the last 90 days.
5. Presence of mental illnesses (registered by psychiatric / mental health facility).
6. Treatment with steroids in the last 30 days (excluding contraceptives and drugs for intranasal and topical administration).
7. Autoimmune diseases or a history of systemic collagenases that require immunosuppressive therapy.
8. Volunteers who have undergone organ transplantation, including bone marrow or peripheral blood stem cell transplants.
9. Immunosuppressive drugs and/or immunomodulators intake for 6 months prior to the start of the Study.
10. Any immunodeficiency (for example, hereditary immunodeficiency, acquired immunodeficiency syndrome [AIDS], etc.).
11. Systolic blood pressure less than 100 mmHg or higher than 139 mmHg; diastolic blood pressure less than 60 mmHg or higher than 90 mmHg; heart rate less than 60 beats / min or more than 100 beats / min.
12. Diabetes mellitus or other forms of glucose tolerance disorders.
13. The medical history of malignant neoplasms, with the exception of basal cell or squamous cell epithelial skin carcinomas, which were removed without any signs of metastasis for 3 years.
14. Blood donation (450 ml or more of blood or plasma) less than 2 months before the start of the Study.
15. Taking narcotic and psychostimulant drugs at the present time or according to the anamnesis.
16. Drinking alcohol above the low-risk level: no more than 20 grams of pure alcohol per day, no more than 5 days a week, alcohol intake within 48 hours before the study drug administration.
17. Smoking: more than 10 cigarettes a day.
18. Planned hospitalization and / or surgical intervention during the period of participation in the Study, as well as 4 weeks before the expected date of study drug administration.
19. Disorders of fat metabolism (pathological hyperlipidemia);
20. Pregnancy or breast-feeding.
21. The presence of a concomitant disease that may affect the evaluation of the Study results or that, in the opinion of the Investigator, will not allow the volunteer to participate in the Study or may affect the conduct of the study and/or its results (including the assessment of safety parameters), any conditions that, in the opinion of the Investigator (doctor), may be a contraindication to participation in the Study.

EXCLUSION CRITERIA

Volunteers will be excluded from the Study in the following cases:

1. Volunteer who does not meet the inclusion criteria and meets at least one exclusion criteria was included in the Study by mistake.
2. Severe violation of the Protocol. The volunteer ignored the Protocol requirements, or the volunteer obtained at least one exclusion criteria during participation in the Study, and further participation causes a risk to the volunteer's health.
3. Follow-up of the volunteer is not possible. The volunteer did not show up for another visit, any attempts to contact the volunteer were unsuccessful. All attempts to contact a volunteer should be documented.
4. Voluntary withdrawal from the Study. A volunteer has the right to withdraw from the Study at any time without providing any reasons. If the volunteer provides such reason, it must be registered with the Case Report Form (CRF).
5. Investigator's decision that the volunteer should be excluded in the interests of the volunteer himself.
6. The development of a serious adverse event before the administration of the study drug.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Occurrence of adverse events (AE) | within 7 days after administration of the study drug
  Occurrence of adverse events (AE) according to CTCAE, v.5.0 (Common Terminology Criteria for Adverse Events).

IPD SHARING:
Plan to Share IPD: No